CLINICAL TRIAL: NCT04907266
Title: Validation Of Chronic Pancreatitis Prognosis Score (COPPS) in a Tropical Cohort of Chronic Pancreatitis
Brief Title: Validation Of Chronic Pancreatitis Prognosis Score (COPPS)
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Kshaunish Das, Professor, Division of Gastroenterology, School of Digestive and Liver Diseases, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: IEC/2018/426
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Structured Questionnaire — A structured proforma to assess outcome

SUMMARY:
Clinical course of chronic pancreatitis is still unpredictable, due to the lack of clinical classification. There is no model to assess disease severity or progression or predict patient outcomes. So we need to validate an objective predictive model - Chronic Pancreatitis Prognosis Score (COPPS) for classification, prognostication and management in Chronic Pancreatitis (CP)

DETAILED DESCRIPTION:
INTRODUCTION Chronic pancreatitis is an inflammatory disease of the pancreas characterized by abdominal pain, repeated episodes of acute pancreatitis, and fibrotic destruction of the organ, resulting in exocrine and endocrine insufficiency. During the last decade, several reports have provided evidence that repeated attacks of acute pancreatitis may progress to chronic pancreatitis [1].

The disease may present clinically either with an individual symptom or a combination of symptoms associated with loss of pancreatic function. The natural history of chronic pancreatitis is usually characterized by progression of tissue damage and various degrees of exocrine and endocrine pancreatic insufficiency, which will become apparent over time, independent of the underlying etiology, chronic pancreatitis evolves toward the same end stage, i.e., pancreatic fibrosis [2].

The prevalence of CP has been approximated at ~50/100,000 population [3]. The underlying etiologies are multifactorial and among many involve excessive alcohol consumption, smoking, genetic predisposition and autoimmune pancreatitis.

It is general knowledge that the terminal stage of chronic pancreatitis results in a loss of organ function, with the clinical manifestations of maldigestion and diabetes mellitus. However, there is little knowledge of the early structural and functional abnormalities because the current diagnostic imaging procedures are not sensitive enough to visualize them and histology is normally not available in these early stages [4].

Abdominal pain is the most frequent symptom of CP. However, the severity, temporal nature, and natural history of pain is highly variable [5].

Chronic pancreatitis encompasses a number of disease entities and can be broadly classified into three forms: chronic calcifying pancreatitis, chronic obstructive pancreatitis, and steroid-responsive pancreatitis (chronic auto immune pancreatitis) [6].

The presentation of multiple clinical symptoms and the frequent occurance of various complications require a well-differentiated therapeutic approach. Current therapies in the management of chronic pancreatitis include conservative measures (analgesics, anti-inflammatory agents, enzyme replacement), endoscopic interventions as well as surgical procedures [7-10] The main reason for the lack of guided strategies in the therapeutic management of chronic pancreatitis is the absence of clearity in the clinically applicable classifications of chronic pancreatitis developed so far, which needs to be developed for guiding management and predicting disease outcome [11].

REVIEW OF LITERATURE For many years, pancreatologists have struggled to achieve a workable classification of chronic pancreatitis. A uniformly accepted and clinically relevant classification is essential to allow for a valid comparison of information among institutions, to improve patient care, and to ensure that patients entered into randomized trials have similar characteristics. Such a classification is also required for staging the disease severity, to plan the management accordingly and to predict disease outcome in both short and long term.

The first classification of chronic pancreatitis was developed at a symposium in Marseilles in 1963, it was based on morphological changes and etiology underlying the disease [12].It correlated clinical features with histology. Pancreatitis was classified as the following four subgroups: acute pancreatitis, relapsing acute pancreatitis, chronic relapsing pancreatitis, and chronic (primarily painless) pancreatitis. The term acute pancreatitis referred to an episode of acute inflammation of the pancreas that resolved completely both clinically and histologically. Relapsing acute pancreatitis referred to recurring episodes of acute pancreatitis that also resolved completely both clinically and histology. The term chronic pancreatitis indicated that histologic changes persisted even after the etiologic agent had been removed. The distinction between chronic relapsing and chronic (primarily painless) pancreatitis was clinical. It was thought that almost all diseases that caused chronic pancreatitis were associated with recurring episodes of pain, and they were therefore termed chronic relapsing pancreatitis, including both chronic pancreatitis caused by alcohol and hereditary pancreatitis. It was recognized that some patients with chronic pancreatitis never experienced pain and that others might experience fewer episodes of pain in time. In summary, at the Marseille Classification Symposium, acute pancreatitis was thought to be associated with complete structural and functional recovery, and it was thought to rarely evolve into chronic pancreatitis. On the other hand, in chronic pancreatitis, structural and functional damage was thought to persist even if the primary cause was eliminated. The major focus of the Marseille Classification of 1963 was pathological anatomy and etiology, and no correlation between anatomical and functional changes was discussed.

It was then generally recognized that reclassification of pancreatitis was required because of the development of new imaging procedures and function tests. At an international workshop in Cambridge in 1983 [13], a revised classification simplified matters by considering pancreatitis as either acute or chronic. Acute pancreatitis was defined as an acute inflammation of the pancreas, usually presenting with abdominal pain and usually associated with increased pancreatic enzymes in the blood or urine. Acute pancreatitis was subdivided into mild and severe cases, and it was recognized that acute pancreatitis could recur. Chronic pancreatitis was defined as an ongoing inflammatory disease typically associated with abdominal pain and characterized by irreversible structural changes and permanent loss of function. It was acknowledged that chronic pancreatitis could recur and was occasionally painless. The Cambridge classification, which was the first clinical grading system for chronic pancreatitis, was based on changes in ductal morphology on endoscopic retrograde pancreatography (ERP) [Table 1] and to some extent had equivalent findings on ultrasound or computed tomography (CT) [14].

Moreover, it was acknowledged that additional studies would be required to provide a grading system of functional impairment. Subsequently, such a grading system of exocrine pancreatic insufficiency has been developed (Table 3) and published [15].

The Cambridge criteria remain the standard for grading of chronic pancreatitis on imaging, but already when it was first introduced, experts stated that morphological changes in chronic pancreatitis might not reflect the functional or histological state of the pancreas and early stages of the disease might be missed [15].

In the revised version of Marseille Classification, published in 1985 [16], the morphological changes that were specified earlier, were linked to a potential loss of endocrine and exocrine organ function. In acute pancreatitis there is a gradation of severity of histologic lesions from mild peripancreatic fat necrosis and interstitial edema to a severe form involving extensive peripancreatic and intrapancreatic fat necrosis, parenchymal necrosis, and bleeding. The process can be localized or diffuse . It was also noted that clinical severity need not correlate with morphological severity. Morphologic characterization of chronic pancreatitis was that of destruction and of permanent loss of exocrine parenchyma in either a focal, segmental, or diffuse pattern, progressive or permanent loss of exocrine or endocrine function, irregular scarring, varying degrees of pancreatic duct dilatation, and preservation of islets of Langerhans. A distinctive form of chronic pancreatitis, obstructive chronic pancreatitis, was also delineated in this re-classification. Descriptive terms that were applied included chronic pancreatitis with focal necrosis, chronic pancreatitis with segmental or diffuse fibrosis, and chronic pancreatitis with or without calculi.

Further modifications in the Marseilles Classification were finally introduced in the consecutively published Marseilles-Rome classification [6]. Two additional forms were introduced- Chronic calcifying pancreatitis and Chronic inflammatory pancreatitis. Chronic inflammatory pancreatitis was characterized by loss of exocrine parenchyma with replacement by diffuse fibrosis with infiltration by mononuclear cells. Chronic calcifying pancreatitis was subdivided into a variety of forms, including hereditary pancreatitis, nutritional pancreatitis (including tropical pancreatitis), and hypercalcemic pancreatitis. They also emphasized on the need for the development of a clinical classification of chronic pancreatitis.

Ammann introduced the concept of stage wise progression in chronic alcoholic pancreatitis. Two stages in the evolution of CP were distinguished: (1) early-stage CP, i.e., no calcification and only minor or no exocrine insufficiency; and (2) late-stage CP, i.e., with calcification and/or persistent exocrine insufficiency. [17] In 2002, Ramesh et al [18] proposed ABC classification which graded chronic pancreatitis based on the presence or absence of clinical pain syndrome and complications like bile duct/ duodenal obstruction/bleeding complications, but it does not clearly differentiate between different degrees of disease severity within a given category, nor does it allow categorization of all possible clinical presentations of chronic pancreatitis.

In 2006, Manchester classification [19] graded chronic pancreatitis into mild, moderate and severe categories. In mild chronic pancreatitis, there was no regular opiate intake (with regular being defined as weekly) and that there be no clinical evidence of impaired pancreatic exocrine or endocrine function or extra-pancreatic complications (duodenal stenosis, portal vein thrombosis and/or distal bile duct stricture). Moderate category has regular abdominal pain requiring opiod use with clinical evidence of impairment of either endocrine or exocrine function without extra-pancreatic complications. End stage chronic pancreatitis has a range of extra-pancreatic complications plus one or more clinical factors to suggest end-stage pancreatic function: either steatorrhoea or diabetes mellitus. [Table 4]

Table 4. MANCHESTER CLASSIFICATION

In 2007, based on the previous chronic pancreatitis classifications, Schneider J et al proposed the MANNHEIM classification [20], grading the disease on the basis of clinical symptoms, imaging findings based on Cambridge classification and pancreatic function insufficiency. It had the following diagnostic criteria-

Definite chronic pancreatitis is established by one or more of the following additional criteria:

1. Pancreatic calcifications
2. Moderate or marked ductal lesions (according to the Cambridge classification)
3. Marked and persistent exocrine insufficiency defined as pancreatic steatorrhea markedly reduced by enzyme supplementation
4. Typical histology of an adequate histological specimen

Probable chronic pancreatitis is established by one or more of the following additional criteria:

1. Mild ductal alterations (according to the Cambridge classification)
2. Recurrent or persistent pseudocysts
3. Pathological test of pancreatic exocrine function (such as fecal elastase-1 test, secretin test, secretin-pancreozymin test)
4. Endocrine insufficiency (i.e., abnormal glucose tolerance test) Borderline chronic pancreatitis is already established and is defined by a typical clinical history of the disease but without any of the additional criteria required for definite or probable chronic pancreatitis. This form is also established as a first episode of acute pancreatitis with or without (1) a family history of pancreatic disease (i.e., other family members with acute pancreatitis or pancreatic cancer) or (2) the presence of risk factors.

   They also proposed a clinical staging system, subcategorizing into an asymptomatic phase (stage 0) and a symptomatic phase (stages I, II, III, IV) of chronic pancreatitis [table 5]. The poorly defined asymptomatic and early phase of chronic pancreatitis, during which clinically recognized symptoms are not present (stage 0 a), was estimated only retrospectively, for example, during surgical intervention or by autopsy. First episode of acute pancreatitis (stage 0 b) was also included since it has been hypothesized that any episode of acute pancreatitis in individuals at risk may cause the later development of chronic pancreatitis. Table 5 . M-ANNHEIM clinical staging of chronic pancreatitis

   This classification also includes a scoring system to determine the severity of the disease to guide clinical treatment decisions and to predict the prognosis of the disease [table 6]. But it is rather a very complex score was not correlated against any valid outcome criteria when first developed [20].

   Table 6. M-ANNHEIM scoring system for the grading of clinical features of chronic pancreatitis In 2009, came the Heidelberg classification [11]which again classified the disease based on clinical features, imaging findings, presence or absence of local complications and end stage disease in the form of exocrine or endocrine insufficiency. Stage A disease was defined as pain of any type and degree and/or attacks of acute pancreatitis, without any complications ; nor steatorrhea, nor insulin-dependent diabetes mellitus. Stage B is the intermediate stage where chronic pancreatitis has led to complications like bile duct obstruction with cholestasis or jaundice ,duodenal obstruction, vascular obstruction , portal/splenic vein hypertension, pancreatic pseudocysts , pancreatic fistula (internal or external), pancreatogenic ascites but clinical exocrine and endocrine function is still preserved. Stage C is the end stage of chronic pancreatitis, where pancreatic fibrosis has led to clinical exocrine and/or endocrine pancreatic function loss (steatorrhea and/or diabetes mellitus). Complications of chronic pancreatitis might or might not be present.

   All these classifications described earlier help to describe the natural progression of the disease by grading the severity on the basis of imaging, clinical symptoms, need for intervention and loss of function, but are neither suited to assess the current severity nor to evaluate short- to mid-term outcomes of the disease [21]. Furthermore, none of the published severity scoring systems have been developed in a prospective cohort of patients nor have they been evaluated for predicting relevant clinical outcome parameters, so in future we need to develop an objective scoring system for classification of chronic pancreatitis which is simple to use on day to day basis yet effective in predicting disease outcome.

   In 2016, Olsen et al did a prospective study in Denmark [22] on their cohort of chronic pancreatitis outpatients and studied various risk factors for the hospitalization rate. On multivariate analysis they demonstrated that high dose opioid treatment (>100 mg per day) and hypoalbuminemia were identified as independent risk factors for hospitalisation.

   Recently in 2017 Bayer et al [21]have developed a simple and dynamic scoring system-Chronic Pancreatitis Prognostic score (COPPS), in a prospective study, comparable to the Turcotte-Child-Pugh-score for liver cirrhosis based on routine laboratory parameters (serum platelet counts, CRP, HbA1c), pain symptoms, body mass index (BMI). They have also validated the same in an independent cohort and found positive co-relation with hospital re-admission rates and duration of hospital stay in the follow up. On this basis they propose that it can be used by general physicians in the outpatient setting and hospitalists alike to reliably predict the risk of hospital (re)admission as a measure of disease severity. This is a new score which need to be further validated in other patient cohort of chronic pancreatitis to prove its utility in predicting disease outcome.

   AIM OF THE STUDY
   * Clinical course of chronic pancreatitis is still unpredictable, due to the lack of clinical classification
   * There is no model to assess disease severity or progression or predict patient outcomes
   * So we need to validate an objective predictive model - Chronic Pancreatitis Prognosis Score (COPPS) for classification, prognostication and management in Chronic Pancreatitis (CP)

   DEFINITION OF CHRONIC PANCREATITIS Diagnosis of chronic pancreatitis was made if one or more met -

   • recurrent bouts of pancreatic pain with documented rise in amylase or lipase activity for a duration of more than one year and radiological evidence (CECT ABDOMEN) supporting the diagnosis
   * pancreatic calcifications and/or MPD dilatation
   * histological proof of chronic pancreatitis
   * unequivocal changes in pancreatic duct morphology
   * Severely abnormal pancreatic function tests with maldigestion [23]

   INCLUSION CRITERIA
   * MEETS THE DEFINITION OF CP
   * Not underwent pancreas related endoscopy/surgery earlier
   * Follow up/index visit in our OPD/ward
   * GIVES INFORMED WRITTEN CONSENT

   EXCLUSION CRITERIA • Pancreatic carcinoma

   OUTCOMES OF THE STUDY PRIMARY OUTCOME
   * Total number of hospitalizations (all reasons)
   * Total number of days spent in hospital within 12 months from inclusion SECONDARY OUTCOME
   * pancreatitis related no of readmissions (episodes of acute pancreatitis, pain episodes , complications, pancreatic endoscopy/sx, infections related to pancreatitis)
   * pancreatitis related complications
   * need for endoscopic or surgical interventions (no. and nature of procedure done)

   MATERIALS AND METHODS

   • Study area: School of Digestive & Liver Diseases, IPGMER and SSKM Hospital, Kolkata.
   * Study population: Patient diagnosed with Chronic Pancreatitis visiting our OPD/Indoors
   * Study Period: June 2018 to December 2019
   * Sample Size: As many patients satisfying inclusion criteria
   * Study Design: Prospective non-randomised Cohort Study.
   * Study area: School of Digestive & Liver Diseases, IPGMER and SSKM Hospital, Kolkata.
   * Study population: Patient diagnosed with Chronic Pancreatitis visiting our OPD/Indoors
   * Study Plan:

     - Enrollment process for 1st 6 months; follow up for 1 year from ENROLLMENT DATE

     - Detailed records will be taken and clinical examination will be carried out as per Proforma designed in each visit

     - All patients will undergo routine blood investigations prospectively from the institute only

     - All the patients will be followed up every 3 monthy - in Pancreatic Clinic or indoor visit or Telephonic
   * Study tool - Structured Questionnaire - Analysis of Previous Medical and Interventional records

     * Blood investigations
   * Statistical Analysis - All continuous variables expressed as MEAN +/- SD - All Categorical data expressed as Proportion/Ratio - Non-parametric statistics, Chi-square test for categorical variables and Kruskal-Wallis test and Dunn´s multiple comparison test for continuous variables.

     * Data entered will be done in MS EXCEL Spread Sheet, Data analysis will be carried out by SPSS version 16.0
     * All P value <0.05 will be considered as statistical significant

   Bibliography

1. Ammann RW, Akovbiantz A, Largiader F, Schueler G. Course and outcome of chronic pancreatitis. Longitudinal study of a mixed medical-surgical series of 245 patients. Gastroenterology 1984;86:820-8.

2. Shrikhande SV, Martignoni ME, Shrikhande M, et al.: Comparison of histological features and inflammatory cell reaction in alcoholic, idiopathic and tropical chronic pancreatitis. Br J Surg 2003, 90:1565-1572 3. Yadav D, Lowenfels AB. The Epidemiology of Pancreatitis and Pancreatic Cancer. Gastroenterology [Internet]. 2013 May [cited 2017 Mar ;144 (6) : 1252-61 4. Nichols MT, Russ PD, Chen YK: Pancreatic imaging: current and emerging technologies. Pancreas 2006, 33:211-20 5. Ammann RW, Muellhaupt B: The natural history of pain in alcoholic chronic pancreatitis. Gastroenterology 1999, 116:1132-40 6. Axon AT, Classen M, Cotton PB, et al. Pancreatography in chronic Pancreatitis: international definitions. Gut 1984;25:1107-1112.

7. Dumonceau JM, Vonlaufen A: Pancreatic endoscopic retrograde cholangiopancreatography (ERCP). Endoscopy 2007, 39:124-30. 8. Dominguez-Munoz JE: Pancreatic enzyme therapy for pancreatic exocrine insufficiency. Curr Gastroenterol Rep 2007, 9:116-22.

9. Van Esch AA, Wilder-Smith OH, Jansen JB, et al.: Pharmacological management of pain in chronic pancreatitis. Dig Liver Dis 2006, 38:518-26. 10. Alexakis N, Halloran C, Raraty M, et al.: Current standards of surgery for pancreatic cancer. Br J Surg 2004, 91:1410-27 11. Büchler MW, Martignoni ME, Friess H, et al. A proposal for a new clinical classification of chronic pancreatitis. BMC Gastroenterol 2009;9:93. 12. Perrier CV. Symposium on the etiology and pathological anatomy of chronic pancreatitis: Marseilles, 1963. Am J Dig Dis 1964;9:371-376. 13. Sarner M, Cotton PB. Classification of pancreatitis. Gut 1984;25:756-759. 14. Banks PA. Classification and diagnosis of chronic pancreatitis. J gastroenterol 2007;42 Suppl 17:148-151.

15. Singer MV, Gyr K, Sarles H. Revised classification of pancreatitis. Report of the Second International Symposium on the Classification of Pancreatitis in Marseille, France, March 28-30, 1984. Gastroenterology 1985;89:683-685.

16. Sarles H, Adler G, Dani R, et al. The pancreatitis classification of Marseilles Rome 1988. Scand J Gastroenterol 1989;24:641-642.

17. Ammann RW. A clinically based classification system for alcoholic chronic pancreatitis: summary of an international workshop on chronic pancreatitis. Pancreas 1997;14:215-221. 18. Ramesh H. Proposal for a new grading system for chronic pancreatitis: the ABC system. J Clin Gastroenterol 2002;35:67-70.

19. Bagul A, Siriwardena AK. Evaluation of the Manchester classification system for chronic pancreatitis. JOP J Pancreas 2006;7:390-396.

20. Schneider A, Löhr JM, Singer MV. The M-ANNHEIM classification of chronic pancreatitis: introduction of a unifying classification system based on a review of previous classifications of the disease. J Gastroenterol 2007;42:101-119 21. Georg Beyer et al. Development and Validation of a Chronic Pancreatitis Prognosis Score in 2 Independent cohorts. Gastroenterology. 2017 Dec;153(6):1544-1554 22. Olesen SS, Poulsen JL, Broberg MCH, et al. Opioid treatment and hypoalbuminemia are associated with increased hospitalisation rates in chronic pancreatitis outpatients. Pancreatol Off J Int Assoc Pancreatol IAP Al 2016 23. Hoffmeister A, Mayerle J, Beglinger C, et al.S3-consensus guidelines on chronic pancreatitis: Definition, aetiology, diagnostic examinations, medical, endoscopic and surgical management of chronic pancreatitis. Z Für Gastro 015;53:1447-1495

ELIGIBILITY:
INCLUSION CRITERIA

* MEETS THE DEFINITION OF CP
* Not underwent pancreas related endoscopy/surgery earlier
* Follow up/index visit in our OPD/ward
* GIVES INFORMED WRITTEN CONSENT

EXCLUSION CRITERIA

* Pancreatic carcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient diagnosed with Chronic Pancreatitis visiting OPD/Indoors
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Total number of hospitalizations (all reasons) | 12 months
  Number of times patient admitted in hospital
Total number of days spent in hospital within 12 months from inclusion | 12 months
  Number of days spent in hospital

SECONDARY OUTCOMES:
pancreatitis related no of readmissions | 12 months
  Admissions due to episodes of acute pancreatitis, pain episodes , complications, pancreatic endoscopy/sx, infections related to pancreatitis
pancreatitis-related complications | 12 months
  Pseudocyst, ascites, biliary stricture, segmental portal hypertension etc.

CONTACTS AND LOCATIONS:
Locations (1):
- IPGMER, Kolkata, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maheshwari A, Patra PS, Ray S, Dhali GK, Das K. External validation of Chronic Pancreatitis Prognosis Score (COPPS): A prospective cohort study. Dig Liver Dis. 2022 May;54(5):654-662. doi: 10.1016/j.dld.2021.08.022. Epub 2021 Sep 17. PMID 34544675